CLINICAL TRIAL: NCT02290002
Title: Calcium Dobesilate Versus Coasting for Prevention of Ovarian Hyperstimulation Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: khalid abd aziz mohamed (Other)
Responsible Party: Sponsor-Investigator, khalid abd aziz mohamed, lecturer of ob/gyn, Benha University
Organization: Benha University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ahmed-khalid 8
Record Dates: First submitted 2014-11-08; First posted 2014-11-13 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Active Comparator): In group A, (Calcium Dobesilate group), 1 cap / 8 hs Calcium Dobesilate ( 500mg) will be given from at day of HCG injection and for 21 days.
  Interventions: Drug: Calcium Dobesilate
- group B (Active Comparator): In group B, coasting (withholding gonadotrophins while maintaining pituitary suppression) for 3 days then either giving triggering or cycle cancellation is done
  Interventions: Other: coasting

INTERVENTIONS:
Drug: Calcium Dobesilate — 1 cap / 8 hs Calcium Dobesilate ( 500mg) will be given at day of HCG injection and for 21 days
  Other Names: doxium
  Arms: group A
Other: coasting — In group B, coasting (withholding gonadotrophins while maintaining pituitary suppression) for 3 days then either giving triggering or cycle cancellation is done
  Arms: group B

SUMMARY:
The purpose of this study is to compare the effect of oral Calcium Dobesilate versus costing in the prevention of ovarian hyperstimulation syndrome (OHSS) in high-risk women underwent intracytoplasmic sperm injection (ICSI).

DETAILED DESCRIPTION:
Two hundred and twenty women at risk of ovarian hyperstimulation syndrome during ICSI cycles will be randomly scheduled into two equal groups. In group A, (Calcium Dobesilate group), 1 cap / 8 hs Doxium ( 500mg) will be given at day of HCG injection and for 3 weeks ; while in group B (Coasting group), coasting (withholding gonadotrophins while maintaining pituitary suppression) follow up every day by measuring E2 for 3 days then either giving triggering or cycle cancellation is done

ELIGIBILITY:
Inclusion Criteria:

* Infertile women undergoing intracytoplasmic sperm injection or polycystic ovarian syndrome (PCO) with one of the following:

  * Presence of more than 20 follicles by ultrasound
  * E2 more than 3000 pg/ml
  * Retrieval of more than 15 follicles

Exclusion Criteria:

* None

Ages: 23 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with ovarian hyperstimulation syndrome (OHSS) | every two weeks for eight weeks
  this will be assessed by:
  Clinically:
  Abdominal bloating Mild abdominal pain Nausea ± vomiting Oliguria Acute respiratory distress syndrome
  By ultrasound Ovarian size usually ˃8 cm Ultrasound evidence of ascites
  Laboratory Haemoconcentration haematocrit ˃45% Hypoproteinaemia

SECONDARY OUTCOMES:
pregnancy rate | 14 days after embryos transfer
  β-hCG (serum hCG test) will be checked 14 days after embryos transfer

CONTACTS AND LOCATIONS:
Overall Officials: ahmed saad, MD, Study Chair — lecturer of ob/gyn; khalid mohamed, MD, Study Director — lecturer of ob/gyn
Locations (1):
- Benha univesity hospital, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: Undecided